CLINICAL TRIAL: NCT05808192
Title: De Novo Metabolic Syndrome in Liver Transplant Patients After Immunosuppression Withdrawal
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Roberta Angelico, Professor, University of Rome Tor Vergata
Other Study IDs: R.S.123.20
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Single Transplant; 5 Years of Follow-up After Transplant, in Which an Attempt Was Made to Suspend IS
Keywords: Metabolic Syndrome, Liver transplantation, Immunosoppression, Tolerance
MeSH Terms: conditions — Metabolic Syndrome | interventions — Immunosuppressive Agents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- tolerant: patients who withdraw IS drugs after LT
  Interventions: Drug: Immunosuppressive
- non tolerant: patients who couldn't wean IS drugs
  Interventions: Drug: Immunosuppressive

INTERVENTIONS:
Drug: Immunosuppressive — compare MS development in patients who achieve to suspend IS drugs after LT and in those who could not suspend.

SUMMARY:
Evaluate de novo onset of metabolic syndrome, NAFLD and NASH in liver transplant recipients who have discontinued immunosuppressive therapy ("tolerant") and in those taking immunosuppressive therapy ("non-tolerant").

DETAILED DESCRIPTION:
A retrospective single-center study was conducted aiming to define the incidence of de novo Metabolic Syndrome (MS) in patients who withdraw Immunosoppression (IS) drugs after Liver Transplant (Tolerant-group) compared to these who couldn't wean IS drugs(non-TOL-group).

ELIGIBILITY:
Inclusion Criteria:

* single LT recipients with an attempt of IS withdrawal
* minimum 5 years follow-up

Exclusion Criteria:

* Liver transplant combined with other organs
* Presence of metabolic syndrome and/or NASH and/or NAFLD as an indication for liver transplantation
* Loss of patient to follow-up

Ages: 49 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 92 patients with liver transplantation who attempted to suspend/ achieve suspension of immunosuppressive therapy, in follow-up in Tor Vergata transplant center.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
relation between MS development and IS in LT recipients | 5 years
  Evaluate the de novo onset of metabolic syndrome, NAFLD and NASH in liver transplant recipients who have discontinued immunosuppressive therapy ("tolerant") and in those who could not withdraw IS ("non-tolerant").

SECONDARY OUTCOMES:
IS withdrawal in LT recipients | 5 years
  Evaluate the clinical course of patients undergoing discontinuation of immunosuppressive therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Roberta Angelico, Rome, Italy